CLINICAL TRIAL: NCT05050669
Title: A Prospective Observational Study to Evaluate Disease Presentation and Progression in Subjects With ENPP1 Deficiency and the Early-Onset Form of ABCC6 Deficiency
Brief Title: Natural History Study of ENPP1 Deficiency and the Early-onset Form of ABCC6 Deficiency
Status: Completed | Type: Observational
Sponsor: Inozyme Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: INZ701-003
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ectonucleotide Pyrophosphatase/phosphodiesterase1 Deficiency; ATP-Binding Cassette Subfamily C Member 6 Deficiency; Generalized Arterial Calcification of Infancy; Autosomal Recessive Hypophosphatemic Rickets
Keywords: ectonucleotide pyrophosphatase/phosphodiesterase 1 deficiency; ENPP1; ATP-binding cassette subfamily C member 6 deficiency; ABCC6; Generalized Arterial Calcification of Infancy; GACI; Autosomal Recessive Hypophosphatemic Rickets Type 2; ARHR2; hypopyrophosphatemia
MeSH Terms: conditions — Arterial calcification of infancy; Hypophosphatemic Rickets, Autosomal Recessive, 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention for this observational study — No Intervention for this observational study

SUMMARY:
The purpose of this prospective study is to characterize the natural history of ENPP1 Deficiency and the early-onset form of ABCC6 Deficiency longitudinally. The study will prospectively gather information about the biochemical, physiological, anatomic, radiographic, and functional manifestations (including patient reported outcomes) of each disease.

DETAILED DESCRIPTION:
Study INZ701-003 is a multicenter, prospective, longitudinal, observational study to evaluate disease presentation, progression, and burden of illness in pediatric subjects aged 2 to <18 years with ENPP1 Deficiency and the early-onset form of ABCC6 Deficiency. Subjects will receive care available at the clinical site along with additional assessments administered by the study team.

To participate in this study, subjects will give informed assent and parents/guardians will provide informed consent.

Subject participation will consist of a Screening Period and an Observation Period.

Assessments will be performed at each visit as indicated in the Schedule of Events.

During the Screening Period, assessments will be performed to determine eligibility.

Screening and Baseline assessments may be conducted on the same day if the Investigator determines that the patient can successfully complete all study procedures in one day due to their age. If not, sites may schedule additional visits, as needed. A subject will be enrolled into the study if they meet all eligibility criteria.

During the Observation Period, subjects will be assessed for changes in their disease in the following areas: measurements of physiological function (including laboratory testing and anatomical and radiographical assessment of calcification and bone mineralization); performance outcomes; patient, caregiver, and physician reported outcomes; and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate must meet all of the following inclusion criteria:

1. Must provide written consent of the legally authorized representative/caregiver and assent for subjects after the nature of the study has been explained and prior to any research-related procedures, following the policies of the clinical site
2. Genetic confirmation of ENPP1 Deficiency or ABCC6 Deficiency
3. Male or female, aged 2 to <18 years
4. In the opinion of the Investigator, must be willing and able to complete all aspects of the study
5. Agree to provide access to relevant medical records

Exclusion Criteria:

Individuals who meet the following exclusion criterion will not be eligible to participate:

1. In the opinion of the Investigator and/or Sponsor, presence of any clinically significant disease (outside of those considered associated with the diagnosis of ENPP1 Deficiency or the early-onset form of ABCC6 Deficiency) that precludes study participation or may confound interpretation of study results, such as an unrelated bone, mineral, or muscle disease or genetic connective tissue disease

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll all eligible subjects aged 2 to <18 years with ENPP1 Deficiency and the early-onset form of ABCC6 Deficiency who consent to participate, with the goal of recruiting up to 20 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Measurement of Plasma Inorganic Pyrophosphate (PPi) in Plasma | Up to 12 months
  For each subject, blood plasma will be assayed for Plasma Inorganic Pyrophosphate (PPi), comparing the subjects baseline value over time
Determination of Arterial Calcification | Up to 12 months
  For each subject, occurrence of arterial calcification will be examined
Determination of Organ Calcification | Up to 12 months
  For each subject, occurrence of organ calcification will be examined
Determination of skeletal radiographs | Up to 12 months
  For each subject, skeletal radiographs will be obtained to determine skeletal abnormalities and will be compared to baseline
Determination of range of motion | Up to 12 months
  For each subject, aged 4 to <18 years, range of motion will be assessed comparing to subjects baseline over time

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — Inozyme Pharma, Inc.
Locations (5):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - CHOP - Robers Center for Pediatric Research, Philadelphia, Pennsylvania
  - Cook Children's Hospital, Fort Worth, Texas
- CHU Sainte-Justine, Montreal, Quebec, Canada
- Royal Manchester University Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided